CLINICAL TRIAL: NCT07060430
Title: Comparison of Kaltenborn Mobilization and Mobilization With Movement (MWM) in Wrist Hypomobility After Colle's Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/76
Record Dates: First submitted 2025-05-28; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Colles Fracture; Hypomobility
MeSH Terms: conditions — Colles' Fracture | interventions — Movement

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kaltenborn mobilization (Experimental): Group 1 will recieve heat therapy and then Kaltenborn mobilization. Supervise exercise protocol will be given Wrist, forearm and fingers ROM and isometric exercises. Introductory hand grip exercises Hand grip strengthening exercises
  Interventions: Procedure: Kaltenborn Mobilization
- Mulligan mobilization with movement (Active Comparator): Group 2 will receive heat therpy and then Mulligan Mobilization with Movement Supervise exercise protocol will be given Wrist, forearm and fingers ROM and isometric exercises. Introductory hand grip exercises Hand grip strengthening exercises
  Interventions: Procedure: Mulligan Mobilization with Movement

INTERVENTIONS:
Procedure: Kaltenborn Mobilization — All participants received a standardized treatment regimen first. This began with the application of a hot pack or infrared therapy for 10 to 15 minutes at the start of each session. then this group will receive Kaltenborn mobilizations with each mobilization technique performed for 10 repetitions, and each repetition maintained for 2 to 3 seconds. Mobilizations included palmar (volar) glide, dorsal glide, radial glide, and ulnar glide. In addition to wrist mobilizations, anterior and posterior glides were applied to the distal radioulnar joint.
  Arms: Kaltenborn mobilization
Procedure: Mulligan Mobilization with Movement — All participants received a standardized treatment regimen first. This began with the application of a hot pack or infrared therapy for 10 to 15 minutes at the start of each session. then this group will receive Mulligan's Mobilization with Movement (MWM) technique, which involved 10 repetitions of each mobilization, with each repetition held for 2 to 3 seconds. First, a lateral glide or rotational movement of the carpal bones on the radius was applied, accompanied by the patient actively performing the intended wrist movement, such as flexion, extension, or deviation. Second, an ulnar-directed mobilization of the radius was provided simultaneously with active patient movement.
  Arms: Mulligan mobilization with movement

SUMMARY:
This study is a randomised control trial and the purpose of this study is to determine comparision of Kaltenborn Mobilization and Mobilization with Movement (MWM) in wrist Hpomobility after Colle's fracture.

DETAILED DESCRIPTION:
Participants will be recruited into their respective groups using a coin toss method. Lower crossed syndrome will be assessed using the following tests:

Kaltenborn mobilization at wrist Mulligan Mobilization with Movement at wrist Wrist, forearm and fingers ROM and isometric exercises. Introductory hand grip exercises Hand grip strengthening exercises

ELIGIBILITY:
Inclusion Criteria:

* Both male and female participants (40-70 years old) Participants who will have diagnosed Colle's fracture and treated conservatively by plaster cast fixation and should referred from department of orthopedic surgery Patients group with post Colle's fractures stiffness

Exclusion Criteria:

* Patients having diagnosed Colle's fracture and treated with invasive procedure like K wiring, ORIF etc.

  * Patient with Neuromuscular injuries.(diagnosed)
  * Rheumatoid arthritis.
  * Patients with metacarpal fracture or compartment syndrome, non-union.(diagnosed)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Range of Motion at wrist | 1st measurement taken before starting session (Baseline measurement) 2nd or post measurement taken after end of sessions (after 3 weeks) (2 points measurement would be taken) 9 treatment sessions in 3 weeks is total time period.
  Range of Motion at wrist will be measured by goniometer
Wrist Pain | 1st measurement taken after 3 or 4 sessions of treatment 2nd or last/post measurement taken at end of session (after 3 weeks) (2 points measurement would be taken).
  Measured by PRWE questionnaire. Patient-Rated Wrist Evaluation is a 15-item questionnaire help to assess wrist pain and disability during daily tasks The Pain Subscale consists of 5 items, ranging from 0 to 10. The total score ranges from 0 (no pain) to 50 (maximum pain).
Functional disability | 1st measurement taken after 3 or 4 sessions of treatment 2nd or last/post measurement taken at end of session (after 3 weeks) 2 points measurement would be taken)
  Measured by PRWE questionnaire. Patient-Rated Wrist Evaluation is a 15-item questionnaire help to assess wrist pain and disability during daily tasks. The Function Subscale includes 10 questions divided into two parts-6 questions assess specific activities, and 4 questions assess usual activities. The score for this subscale also ranges from 0 (no difficulty) to 50 (maximum difficulty).

SECONDARY OUTCOMES:
Grip Strength | 1st measurement taken before starting session (Baseline measurement) 2nd or post measurement taken after end of sessions (after 3 weeks) (2 points measurement would be taken) 9 treatment sessions in 3 weeks is total time period.
  Hand held dynamometer was used to assess patient's grip strength. To assess strength, the person sat on chair with 90-degree hip and knee flexion, shoulder in adduction, and elbow flexed to 90 degrees. The forearm and wrist were in a resting position. The dynamometer is placed in the person's hand, and the therapist or examiner gently supports the base of the device. The person was asked to clench the dynamometer as hard as they can for a few seconds, maintaining a smooth and consistent effort. The dynamometer displayed the force generated by the person's grip, and the reading was recorded. The process was usually repeated multiple times (e.g., three trials) to get an average reading and ensure reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan